CLINICAL TRIAL: NCT04837027
Title: Balance Versus Aerobic Training in Degenerative Cerebellar Diseases
Brief Title: Effect of Training on Brain Volume in Ataxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAT1306
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Spinocerebellar Ataxias
Keywords: Ataxia; Cerebellum; Cerebellar degeneration
MeSH Terms: conditions — Spinocerebellar Ataxias; Ataxia

STUDY DESIGN:
Intervention Model Description: Single blinded randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will know that the participant has received balance or aerobic training, but will not be aware of which group the participant belonged.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic training (Experimental): Participants will be given a stationary exercise bike for home use. They will be instructed to use the exercise bike five times a week for thirty-minute sessions. The exercise intensity prescription will be based on the subject's VO2max determined on pre-test day. The exercise program will start at 60% of intensity per session, and then will be increased by steps of 5% intensity every 2 sessions until participants reach 30 minutes of training at 80% intensity. Participants will be contacted weekly by e-mail or phone to answer any questions about the exercise protocol and will be instructed to log each training session. Subjects will record duration of exercise, perceived exertion, average heart rate, maximum heart rate, and distance.
  Interventions: Behavioral: Aerobic training
- Balance training (Active Comparator): Balance Training A physical therapist will tailor a home balance training program for each participant based on pre- training capabilities. Subjects will be asked to perform exercises five times a week for thirty-minute sessions. Both dynamic and static exercises will be performed in sitting and standing positions. Exercises will start with stabilizing in a challenging static position and progress to dynamic arm and leg movements in the same or modified position. Participants will be contacted weekly by e-mail or phone to answer any questions about the exercise protocol and will be required to log their exercise effort in terms of frequency and level of balance challenge. Individuals will be instructed to perform more difficult exercises if balance
  Interventions: Behavioral: Balance training

INTERVENTIONS:
Behavioral: Aerobic training — Aerobic training on stationary bike 5x a week for 30 minutes a day
  Arms: Aerobic training
Behavioral: Balance training — Training 5x a week for 30 minutes. Standard of care
  Arms: Balance training

SUMMARY:
The primary aim is to show balance training improves DCD individual's ability to compensate for their activity limitations, but does not impact disease progression.

The second aim is to demonstrate aerobic exercise improves balance and gait in DCD persons by affecting brain processes and slowing cerebellar atrophy.

DETAILED DESCRIPTION:
Individuals with degenerative cerebellar disease (DCD) exhibit gradual loss of coordination resulting in impaired balance, gait deviations, and severe, progressive disability. With no available disease-modifying medications, balance training is the primary treatment option to improve motor skills and functional performance. There is no evidence, however, that balance training impacts DCD at the tissue level.

Aerobic training, on the other hand, may modify DCD progression as evident from animal data. Compared to sedentary controls, aerobically trained DCD rats have enhanced lifespan, motor function, and cerebellar Purkinje cell survival. Numerous animal studies also document that aerobic training has a direct, favorable effect on the brain that includes production of neurotrophic hormones, enhancement of neuroplasticity mechanisms, and protection from neurotoxins.

The effects of aerobic training in humans with DCD are relatively unknown, despite these encouraging animal data. A single study to date has evaluated the benefits of aerobic exercise on DCD in humans, and this was a secondary outcome of the study. Although participants performed limited aerobic training during the study, modest functional benefits were still detected.

The main objective of this project will be to compare the benefits of aerobic versus balance training in DCD. We hypothesize that both aerobic and balance training will improve function in DCD subjects, but that the mechanisms in which these improvements occur differ. 1) Balance training improves DCD individual's ability to compensate for their activity limitations, but does not impact disease progression. 2) Aerobic exercise improves balance and gait in DCD persons by impacting the cerebellum

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with spinocerebellar ataxia

  * Cerebellar atrophy on MRI
  * Prevalence of ataxia on clinical exam
  * Ability to safely ride a stationary exercise bike

Exclusion Criteria:

* Other neurologic conditions • Heart disease

  * Cognitive impairment
  * Medical instability

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

PRIMARY OUTCOMES:
Cerebellar volume | 6 months
  Cranial MRI will be performed in all participants using a 3-T scanner. Using each individual's T1-weighted image, structural imaging measures of cerebellar brain volume will be derived using the FreeSurfer software package (http:// surfer.nmr.mgh.harvard.edu/). FreeSurfer will automatically assign a neuroanatomic label to each voxel. From this labeling, a set of volumetric regions of interest is defined. The calculated volume within the cerebellar region is adjusted for variations in individual's intracranial brain volume (ICV) which is measured using BrainWash (an automatic
  - Page 3 of 5 [DRAFT] -
  multi-atlas skull-striping software package). We will process the longitudinal T1-weighted images

SECONDARY OUTCOMES:
Cognition | 6 months
  The NIH toolbox will be used before and after training to determine impact of training on cognition
Ataxia severity | 6 months
  The Scale for the Assessment and Rating of Ataxia (SARA) will be done to before and after training. This scale ranges from 0 to 40 with higher scores indicating more ataxia
Gait speed | 6 months
  Participants will walk 8 meters as fast as possible
Balance | 6 months
  The dynamic gait index will be performed to test balance

CONTACTS AND LOCATIONS:
Overall Officials: Scott Barbuto, MD PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No